CLINICAL TRIAL: NCT06351605
Title: A Multi-Center Registry Study to Assess the Safety and Effectiveness of Photobiomodulation in Participants With Dry Age-Related Macular Degeneration (EUROLIGHT)
Brief Title: A Registry Study to Assess Photobiomodulation in Dry Age-Related Macular Degeneration (EUROLIGHT) (EUROLIGHT)
Status: Recruiting | Type: Observational
Sponsor: LumiThera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP006
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Dry Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Photobiomodulation (PBM): Valeda Light Delivery System The Valeda Light Delivery System will deliver two alternating and sequential treatments of 590 nm and 850 nm for 35 seconds, or a total of 70 seconds; and 660 nm for 90 seconds, or a total of 180 seconds.
  Interventions: Device: Valeda Light Delivery System

INTERVENTIONS:
Device: Valeda Light Delivery System — The Valeda Light Delivery System will deliver two alternating and sequential treatments of 590 nm and 850 nm for 35 seconds, or a total of 70 seconds; and 660 nm for 90 seconds, or a total of 180 seconds.

SUMMARY:
The EUROLIGHT study is being conducted to collect real life data for the safety and effectiveness of PBM in dry AMD, in routine clinical practice both retrospectively and prospectively.

DETAILED DESCRIPTION:
This is a multi-center, retrospective and prospective registry study on the use of the Valeda® PBM system as a treatment for visual improvement in participants with dry AMD. The target is at least 25 participants/site in up to 20 participating sites in Europe.

Participants will or will have received nine non-invasive, short treatments over three to four weeks starting at Baseline (BL), with up to five additional rounds of treatment every four to six months, or as determined by the Investigator.

Standard visual outcome measurements collected will include visual acuity (either ETDRS BCVA or LogMAR) prior to and following treatment. OCT and Fundus Autofluorescence (FAF) imaging of the retina should be taken at screening, and after each round of treatment. As this is a registry study, missing

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis or confirmation of diagnosis of dry AMD disease by Investigator
2. Able to communicate well with the Investigator and able to understand and comply with the requirements of the study
3. Informed of the nature of this study and has provided written, informed consent (participants enrolled retrospectively will need to be contacted and sign an informed consent form prior to their data being used).

Exclusion Criteria:

1. Signs of active, inactive or history of exudative macular neovascularization (MNV)
2. History or active accumulation of intra and subretinal fluid of any cause (e.g., diabetic macular oedema, central serous retinopathy, cystoid macular oedema)
3. Use of any photosensitizing agent (e.g. topicals, injectables) activated by the Valeda Light Deliver System within 30 days prior to treatment without consulting participant's physician
4. Has any known photosensitivity to yellow light, red light, or near infrared radiation (NIR), or has a history of light activated CNS disorders (e.g. epilepsy, migraine)
5. In the opinion of the Investigator, is unlikely to comply with the study protocol or has a history or current evidence of any condition that, in the opinion of the investigator, might interfere with the participant's involvement in the trial, or is not in the best interest of the participant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient population for this study will consist of a target of at least 25 male and female participants per site of any ethnic background and with a diagnosis of dry AMD by the Investigator or confirmed by the Investigator. The participant must meet all the inclusion criteria, have none of the exclusion criteria, and give their written Informed Consent to participate in this clinical study.
  Only if the participant is interested in participating, s/he would be given the option to sign the study consent and start the study procedures, or if retrospectively signing the informed consent form, have their data used in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) | 31 months
  Mean change from baseline in BCVA.

SECONDARY OUTCOMES:
OCT Imaging | 31 months
  OCT instruments will be used to image the retina for diagnosis and anatomical assessments (general retinal thickness and drusen volume) of dry AMD pathology
FAF Imaging | 31 months
  FAF is used to evaluate both hypoautofluorescence (GA) and hyperauto-fluorescence and drusen byproducts, the deposition of lipofuscin in the retinal pigment epithelium D3001-CSP006 14MAY2023 V2.0 CONFIDENTIAL Page 22 of 42 (RPE).

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Croissant, MBA, Study Director — LumiThera, Inc.
Locations (1):
- Oslo University Hospital, Oslo, Norway